CLINICAL TRIAL: NCT05401786
Title: Anti-PD-1 Re-challenge After Immune Priming by Ipilimumab and Immune Boosting by Radiotherapy in Advanced NSCLC
Acronym: RAD-IO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M21RAD
Record Dates: First submitted 2022-05-17; First posted 2022-06-02 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab; cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-CTLA-4, SBRT and PD1 (Experimental): Participants will receive 1 dose of ipilimumab (1mg/kg intravenously) on day 1. After 1 week the participants will receive SBRT (3x8Gy) on at least 1 but no more than 4 tumor lesions.
  Within 1 week of the last radiation fraction participants will start with cemiplimab (350mg intravenously every 3 weeks) until disease progression, unacceptable toxicity, patient request for discontinuation, or up to 2 years of treatment
  Interventions: Drug: Ipilimumab; Drug: Cemiplimab; Radiation: SBRT

INTERVENTIONS:
Drug: Ipilimumab — Anti-CTLA-4
Drug: Cemiplimab — PD-1 inhibition
Radiation: SBRT — Stereotactic Body Radiotherapy

SUMMARY:
Still many advanced non-small cell lung cancer (NSCLC) patients do not benefit from PD-(L)1 inhibition or will eventually develop progression through secondary resistance. Inhibition of CTLA-4, application of radiotherapy together with PD-1 inhibition showed synergistic effects and is deemed safe.

DETAILED DESCRIPTION:
Still many advanced non-small cell lung cancer (NSCLC) patients do not benefit from PD-(L)1 inhibition or will eventually develop progression through secondary resistance. The aim of this study is to investigate whether the combining of T cell priming by CTLA-4 inhibition (ipilimumab) ad subsequent immune boosting by stereotactic body radiotherapy (SBRT) on 1-4 tumor lesions can re-invigorate the response on PD-1 inhibition (cemiplimab) after initial non-response or secondary resistance to anti-PD-(L)1 treatment. Elaborate translational research by repeat biopsies in combination with blood collection during the different stages of treatment will help improve understanding of the joint effort of these different interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Have proven diagnosis of recurrent advanced NSCLC, irrespective of histological subtype.
2. Be willing and able to provide written informed consent/assent for the trial.
3. Must still have measurable disease based on RECIST 1.1 after application of study SBRT. Lesions that were irradiated prior to the study, but have progressed since irradiation but prior to study inclusion will be allowed as measurable disease.
4. Must provide newly obtained tissue from a core or excisional biopsy of a tumor lesion and are willing to have a second biopsy performed from any non-irradiated lesion after the radiation and immune-modulating treatment. This lesion may be used for RECIST measurements.
5. Have a performance status of 0 or 1 on the ECOG Performance Scale.
6. Stage IV NSCLC treated with at least PD-(L)1 blockade. There is no maximum number of previous lines of systemic treatment. Patients with both primary or acquired resistance to PD-(L)1 inhibition may be considered eligible. However, in the 1st stage ≥4 of 12 patients, in the 2nd stage a total of ≥8 of 25 patients and in the 3rd stage a total of ≥27 of 54 patients need to fulfill the definition of acquired resistance. Also, a maximum of 27 patients with a PD-L1 negative tumor will be included.
7. Have at least 2 separate (metastatic) lesions of which one is eligible for irradiation and another for biopsy and RECIST tumor evaluation.
8. Demonstrate adequate organ function. All screening labs should be performed within 14 days of treatment initiation.
9. Female subject of childbearing potential should have a negative serum pregnancy test within 72 hours prior to receiving the 1st dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 6 months after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
11. Male subjects should agree to use an adequate method of contraception starting with the 1st dose of study therapy through 6 months after the last dose of study therapy

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Has a non-smoking-related targetable driver mutation, e.g. EGFR, ALK, RET or ROS1. Patients with advanced NSCLC with a smoking-related targetable driver mutation, e.g. KRAS or BRAF, may be found eligible if they have a history of ≥10 PY, but only when all options for targeted therapy have been exhausted and when progression on previous PD-(L)1 blockade has occurred.
2. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the 1st dose of treatment.
3. Has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: Patients who experienced significant autoimmune side effects related to previous PD-(L)1 checkpoint inhibition, i.e. requiring use of steroids or other anti-inflammatory drugs and/or the need to (temporarily) withhold PD-(L)1 checkpoint inhibition, may be considered eligible after discussion with the coordinating investigator if adverse events have recovered, i.e. ≤ Grade 1 or at baseline.
   * Note: If subjects received major surgery (defined as surgical intervention requiring general or spinal anesthesia and hospital admission), they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy. Major surgery within 14 days prior to start of study treatment is not allowed.
4. Has had previous radical radiation to any tumor site within 3 months prior to study Day 1. Previous palliative radiation to any tumor site is not considered an exclusion criterion; however, this site will not be eligible for SBRT, biopsy location or RECIST tumor evaluation within this study.
5. Has received prior therapy with any antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways other than PD-(L)1 blockade, e.g. anti-CD137 or a CTLA-4 antibody.
6. Patients who have uncontrolled central nervous system (CNS) metastases. Patients who have untreated asymptomatic CNS metastases no greater than 2cm before start of treatment may be eligible. Patients who have any CNS lesion that is symptomatic, greater than 2cm, show significant surrounding edema on MRI scan or have leptomeningeal disease will not be eligible. Patients who have previously been treated for CNS metastases are eligible when they comply with the hereby mentioned criteria.

   NB. A brain lesion is not amendable for study SBRT.
7. Has a known additional malignancy that is progressing or requires active treatment.
8. Has an active autoimmune disease or a documented history of clinically severe autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Subjects who require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Patients with an active or history of autoimmune disease or syndrome who underwent previous PD-(L)1 checkpoint inhibition without significant side effects, i.e. not requiring use of steroids or other anti-inflammatory drugs and/or the need to (temporarily) withhold PD-(L)1 checkpoint inhibition, may be considered eligible for this trial after discussion with the coordinating investigator. Requirement for immunosuppressive doses of systemic corticosteroids ≤10 mg/day prednisone or equivalent may be considered eligible after discussion as well.
9. Has evidence of symptomatic interstitial lung disease or an active, non-infectious pneumonitis.
10. Has an active infection requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Rate | Through study completion, an average of 1 year
  Number of participants with complete response or partial response within the first 6 months or stable disease lasting for minimum 6 months

SECONDARY OUTCOMES:
Objective Response Rate | 12 weeks after re-introduction of PD-1 inhibition (day 1 of week 15)
  Number of participants with complete response or partial response
Disease Control Rate | 12 weeks after re-introduction of PD-1 inhibition (day 1 of week 15)
  Number of participants with complete response, partial response, or stable disease
Best overall response | Through study completion, an average of 1 year
  Best overall response at any time point
Progression Free Survival | From date of start of treatment until first documented progression or the date of death assessed up to 100 months
  Time between start of treatment and progressive disease or death
Overall Survival | From date of start of treatment until the date of death assessed up to 100 months
  Time between start of treatment and death
Safety of the study procedure | Up to 90 days after last study drug intake
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

OTHER OUTCOMES:
Genetic characteristics and signatures of responders vs non-responders 1 | At baseline and week 3 (before initiation of PD-1 inhibition)
  Whole Exome Sequencing of tumor biopsies
Genetic characteristics and signatures of responders vs non-responders 2 | At baseline and week 3 (before initiation of PD-1 inhibition)
  RNA sequencing of tumor biopsies
Changes in TCR repertoire | At baseline and week 3 (before initiation of PD-1 inhibition)
  Changes in TCR repertoire at baseline versus on-treatment tumor biopsies
Changes in protein expression | At baseline and week 3 (before initiation of PD-1 inhibition)
  Multi-staining immunohistochemistry analysis at baseline versus on-treatment tumor biopsies
Changes in blood proteomics profile | At baseline, week 2, 3 and 5 on treatment and at end-of-treatment (an average of 1 year)
  Changes in blood proteomics profile during treatment
Changes in ctDNA | At baseline, week 2, 3 and 5 on treatment and at end-of-treatment (an average of 1 year)
  Changes in ctDNA during treatment

CONTACTS AND LOCATIONS:
Overall Officials: W.S.M.E Theelen, MD,PhD, Principal Investigator — NKI-AvL
Locations (1):
- Antoni van Leeuwenhoek - Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided